CLINICAL TRIAL: NCT00435812
Title: A Phase III Safety and Efficacy Study to Compare Immune Responses Following Injection With Either Two Doses of HEPLISAV™ or Three Doses of Engerix-B®
Brief Title: Safety and Efficacy of HEPLISAV™ Hepatitis B Virus Vaccine Compared With Engerix-B® Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DV2-HBV-10; 2006-006743-31 (EudraCT Number)
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis B
Keywords: HBV vaccine; Hepatitis B vaccine; Hepatitis B; Hepatitis; HBV; Immunostimulatory sequence (ISS)
MeSH Terms: conditions — Hepatitis B; Hepatitis | interventions — Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HEPLISAV and/or Placebo (Experimental): 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018)
  Interventions: Biological: HEPLISAV and/or Placebo
- Engerix-B (Active Comparator): 1.0 mL Engerix-B
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: HEPLISAV and/or Placebo — Intramuscular (IM) injections on Week 0, Week 4; placebo (saline) injection at Week 24
  Other Names: HEPLISAV; Hepatitis B vaccine (recombinant), adjuvanted
  Arms: HEPLISAV and/or Placebo
Biological: Engerix-B — Intramuscular (IM) injections on Week 0, Week 4, and Week 24
  Other Names: Hepatitis B vaccine (recombinant)
  Arms: Engerix-B

SUMMARY:
The purpose of this study is to find out if a new investigational hepatitis B virus vaccine, HEPLISAV™, is safe and effective compared with Engerix-B® vaccine in subjects 11-55 years old. The primary hypothesis is that the seroprotective immune response of HEPLISAV™ is at least as good as that of Engerix-B®.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of two injections of HEPLISAV™, compared with three injections of a commercially available hepatitis B virus (HBV) vaccine, Engerix-B®, in subjects 11 to 55 years old. About 2,400 subjects will be included in the study. Once subjects are consented, screened, and randomized to treatment, all subjects will receive a total of three injections over a 24-week period, with a follow-up visit at 28 weeks. Subjects randomized to Engerix-B® will receive 3 injections of active vaccine, while subjects randomized to HEPLISAV™ will receive 2 injections of active vaccine plus 1 injection of placebo. Safety and tolerability will be evaluated by occurrence of adverse events, periodic laboratory tests, vital signs, and local/systemic reactogenicity.

Comparison: Subjects will receive treatment with either HEPLISAV™ or the comparator vaccine, Engerix-B®.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Is serum negative for HBV antibodies

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Any previous HBV infection
* Previous vaccination with any HBV vaccine (1 or more doses)
* Any autoimmune disease
* Received any blood products or antibodies within 3 months prior to study entry
* Ever received an injection with DNA plasmids or oligonucleotides
* Received any vaccines within 4 weeks prior to study entry
* Received any other investigational medicinal agent within 4 weeks prior to study entry

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2428 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Tyler Martin, Sr, MD, Study Director — Dynavax Technologies Corporation
Locations (18):
- Canada (12):
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Winnipeg, Manitoba
  - Mount Pearl, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Ottawa, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Charlottetown, Prince Edward Island
  - Montreal, Quebec
  - Québec, Quebec
- Germany (6):
  - Berlin
  - Hamburg
  - Leipzig
  - Magdeburg
  - Munich
  - Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Dynavax Webpage — http://www.dynavax.com

RESULTS

PARTICIPANT FLOW:
Groups:
- HEPLISAV and/or Placebo: 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018)
  HEPLISAV and/or Placebo: Intramuscular (IM) injections at Week 0 and Week 4, plus a placebo (saline) injection at Week 24
Period: Overall Study
Arm/Group | HEPLISAV and/or Placebo | Engerix-B
Started | 1820 | 608
Completed | 1757 | 590
Not Completed | 63 | 18

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population: All participants who received at least 1 study injection and had any post-baseline safety data.
  NOTE: One (1) subject randomized to the Engerix-B group received HEPLISAV in error and was analyzed in the HEPLSAV group for the Safety Analysis Population
Groups:
- HEPLISAV and/or Placebo: 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018) HEPLISAV and/or Placebo: Intramuscular (IM) injections at Week 0, Week 4, plus a placebo (saline) injection at Week 24
- Total: Total of all reporting groups
Arm/Group | HEPLISAV and/or Placebo | Engerix-B | Total
Number analyzed (Participants) | 1821 | 607 | 2428
Age, Customized [Count of Participants; unit: Participants]
  11 to 17 years | 11 | 2 | 13
  ≥18 and ≤ 55 years | 1810 | 605 | 2415
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 959 | 346 | 1305
  Male | 862 | 261 | 1123
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1123 | 366 | 1489
  Germany | 698 | 241 | 939

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Seroprotective Immune Response
Description: Percentage of subjects who have a seroprotective immune response (anti-HBsAg ≥ 10 milli-international unit (mIU)/mL) after the final active injection in each treatment group (Week 12 for HEPLISAV™ and Week 28 for Engerix-B®)
Time Frame: Week 12 for HEPLISAV and Week 28 for Engerix-B
Population: Per Protocol Population: Subjects who met eligibility criteria, did not violate the protocol in a substantial manner, received all protocol-specified study injections, had their primary serology and all injections within the specified day ranges, and had serology at their primary endpoint (Week 12 for HEPLISAV group and Week 28 for Engerix-B group)
Measure: Number; unit: Percentage of Participants
Arm/Group | HEPLISAV and/or Placebo | Engerix-B
Number analyzed (Participants) | 1520 | 523
Percentage of Participants | 95.1 | 81.3

2. Secondary Outcome: Percentage of Participants With Local and Systemic Reactions to Injections
Time Frame: Within 7 days post-injection for Post Injection Reactions
Population: Safety Analysis Population: All participants who received at least 1 study injection and had any post-baseline data.
Measure: Number; unit: Percentage of subjects
Arm/Group | HEPLISAV and/or Placebo | Engerix-B
Number analyzed (Participants) | 1821 | 607
Percentage of subjects
  Local Reaction : Injection 1 | 40.4 | 34.1
  Local Reaction : Injection 2 | 35.8 | 24.8
  Local Reaction : Injection 3 | 6.5 | 20.5
  Systemic Reaction : Injection 1 | 27.1 | 29.2
  Systemic Reaction : Injection 2 | 21.2 | 18.5
  Systemic Reaction : Injection 3 | 12.8 | 14.7

ADVERSE EVENTS:
Description: Adverse events were assessed for safety analysis population: All participants who received at least 1 study injection and had any post-baseline safety data
Arm/Group | HEPLISAV and/or Placebo | Engerix-B
Serious Adverse Events (participants affected / at risk) | 28/1821 | 13/607
Other Adverse Events (participants affected / at risk) | 602/1821 | 191/607
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV and/or Placebo (N=1821) | Engerix-B (N=607)
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Salpingo-oophoritis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Guillain-barre syndrome (Nervous system disorders) | 1 | 0
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Granulomatosis with polyangiitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV and/or Placebo (N=1821) | Engerix-B (N=607)
Nasopharyngitis (Infections and infestations) | 303 | 100
Back pain (Musculoskeletal and connective tissue disorders) | 94 | 29
Headache (Nervous system disorders) | 205 | 62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less